CLINICAL TRIAL: NCT02045212
Title: A Preliminary Double Blind Clinical Study, Efficacy Study of RPh201 Treatment of Ischemic Optic Neuropathy (ION).
Brief Title: Safety and Efficacy Study of RPh201 Treatment of Ischemic Optic Neuropathy (ION).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regenera Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGN-ON-001
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Non-arteritic Ischemic Optic Neuropathy; Optic Nerve Injuries
Keywords: Ischemic Optic Neuropathy; Traumatic Neuropathy; Non Arteritic Ischemic Neuropathy (NAION)
MeSH Terms: conditions — Optic Nerve Injuries; Optic Neuropathy, Ischemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RPh201 (Experimental): 3/6 month treatment schedule, consisting of bi-weekly SC administration of the RPh201
  Interventions: Drug: RPh201
- Placebo (Placebo Comparator): 3/6 month treatment schedule, consisting of bi-weekly SC administration of the Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPh201 — SC injection twice a week during 13/26 weeks
  Arms: RPh201
Drug: Placebo — SC injection twice a week during 13/26 weeks
  Arms: Placebo

SUMMARY:
The study objectives are to assess any changes in visual acuity and visual field observed following the administration of RPh201 during an overall treatment period of at least 13 consecutive weeks with an option to extended the treatment phase to another 13 weeks (26 weeks total), and at the follow-up visit at 3 month after end of treatment in patients with optic nerve neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants, either men or women are ≥ 18 years of age.
2. Diagnosis of ischemic optic neuropathy unilateral or bilateral:

   1. Traumatic Neuropathy
   2. Ischemic optic neuropathy - Non Arteritic Ischemic Neuropathy (NAION)
3. Corrected Visual acuity equal or worse than 6/60 or visual field of less than 15 degrees or both.
4. Field of view with a reduction from 10 degrees to one quarter situations functions.
5. Participant understands the nature of the procedure and provides written informed consent prior to any study procedure.
6. Women of child bearing potential must use adequate birth-control precautions.

Exclusion Criteria:

1. Glaucoma
2. Neuropathy caused by tumors.
3. Neuropathy caused by infections
4. Mitochondrial optic neuropathies
5. Nutritional, Radiation, Toxic optic neuropathies
6. Retinal diabetic complications
7. Hereditary optic neuropathies
8. Patients with complete SCOTOMA beyond three quarters.
9. Clinical evidence for presence of infection.
10. Patient is receiving, or has received within one month prior to enrollment corticosteroids, immunosuppressive drugs, cytotoxic agents, radiation therapy and chemotherapy.
11. Patient has a history of alcohol or drug abuse within the last two years.
12. Female patients who are pregnant or nursing, or of childbearing potential and are not using adequate contraception.
13. Participation in another clinical trial within 60 days prior to the Screening Visit or during this study.
14. Clinically significant and/or uncontrolled condition or other significant medical disease
15. Clinically significant uncontrolled retinal disease (AMD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Segal,, MD, Principal Investigator — Head of the Ophthalmology Department, Western Galilee-Nahariya Medical Center Nahariya, Israel
Locations (1):
- Ophthalmology Department, Western Galilee-Nahariya Medical Center, Nahariya, Israel

REFERENCES:
- [Background] Rath EZ, Hazan Z, Adamsky K, Solomon A, Segal ZI, Levin LA. Randomized Controlled Phase 2a Study of RPh201 in Previous Nonarteritic Anterior Ischemic Optic Neuropathy. J Neuroophthalmol. 2019 Sep;39(3):291-298. doi: 10.1097/WNO.0000000000000786. PMID 31430268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RPh201 | Placebo
Started | 13 | 9
Completed | 11 | 8
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Finished 13 weeks, chose not to extend | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPh201 | Placebo | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.46 (8.1) | 60.33 (5.8) | 61.00 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Israel | 13 | 9 | 22
Height [Mean (Standard Deviation); unit: metres] | 1.7 (0.12) | 1.7 (0.12) | 1.7 (0.12)
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (13.58) | 95.5 (24.54) | 88.0 (19.38)
BMI [Mean (Standard Deviation); unit: kg per metre squared] | 29.16 (4.24) | 34.77 (5.52) | 31.46 (5.46)

OUTCOME MEASURES:

1. Primary Outcome: Mean Increase From Baseline in ETDRS Letters Read at 26 Weeks and Off-drug Follow-up Visit
Description: Best Corrected Visual Acuity (BCVA) was assessed at all the visits, with refraction as necessary. VA measurements were taken in a sitting position at a test distance of 4 meters using early treatment diabetic retinopathy study (ETDRS) charts.
Time Frame: 26/39 weeks
Population: Efficacy
Measure: Mean (Standard Error); unit: EDTRS Letters
Arm/Group | RPh201 | Placebo
Number analyzed (Participants) | 12 | 8
EDTRS Letters
  Changes in BCVA from baseline to week 26: number analyzed (Participants) | 11 | 8
  Changes in BCVA from baseline to week 26 | 15 (4.6) | 7 (5.4)
  changes in BCVA from baseline to 39 weeks | 9 (5.6) | 6 (4.7)

2. Secondary Outcome: Number of Participants With Adverse Events Assessed by Vital Signs, Clinical Laboratory and Physical Exam
Description: Safety and tolerability multiple ascending SC doses as assessed by adverse events, vital signs, clinical laboratory and physical exam
Time Frame: 26/39 weeks
Measure: Number; unit: participants
Groups:
- RPh201: 26 weeks treatment schedule, consisting of bi-weekly SC administration of the RPh201
  RPh201: SC injection twice a week during 26 weeks
- Placebo: 26 weeks treatment schedule, consisting of bi-weekly SC administration of the Placebo
  Placebo: SC injection twice a week during 26 weeks
Arm/Group | RPh201 | Placebo
Number analyzed (Participants) | 13 | 9
participants
  Visual acuity ocular safety in fellow eye | 0 | 1
  Visual field ocular safety in fellow eye | 0 | 1

3. Primary Outcome: Changes in Visual Field Observed Following the Treatment
Description: Visual field mean deviation (MD) changes from the screening at week 26 using with the HVF 24-2 FASTPAC program using the size III or Size V test stimulus
Time Frame: 26 weeks
Population: Efficacy
Measure: Mean (Standard Error); unit: dB
Groups:
- RPh201: 26 weeks treatment schedule, consisting of bi-weekly SC administration of the RPh201
  RPh201: SC injection twice a week during up to 26 weeks
- Placebo: 26 weeks treatment schedule, consisting of bi-weekly SC administration of the Placebo
  Placebo: SC injection twice a week during up to 26 weeks
Arm/Group | RPh201 | Placebo
Number analyzed (Participants) | 11 | 8
dB
  Changes Visual Field size III: number analyzed (Participants) | 3 | 4
  Changes Visual Field size III | 7.85 (5.8) | 0.84 (1.47)
  Changes Visual Field size V: number analyzed (Participants) | 8 | 4
  Changes Visual Field size V | 0.41 (1.66) | 0.49 (2.59)

4. Primary Outcome: Changes Mean RNFL Thickness in NAION Eyes Change From Screening to Week 26
Description: TMean RNFL thickness measured by OCT. The data are in microns, as measured with an Opko OCT machine.
Time Frame: 26 weeks
Population: Efficacy
Measure: Mean (Standard Error); unit: µm
Arm/Group | RPh201 | Placebo
Number analyzed (Participants) | 11 | 8
µm | -4.6 (1.58) | -1.8 (2.08)

ADVERSE EVENTS:
Arm/Group | RPh201 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/13 | 1/9
Other Adverse Events (participants affected / at risk) | 13/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPh201 (N=13) | Placebo (N=9)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Visual acuity decreased (Eye disorders) | 1 (1) | 0 (0)
Brucellosis (Infections and infestations) | 1 (1) | 0 (0)
Ischemic optic neuropathy - AION right eye (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPh201 (N=13) | Placebo (N=9)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 4 (5) | 0 (0)
Conjunctival irratation (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Corneal defect (Eye disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 2 (2) | 2 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye Movement Disorder (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 2 (2)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 2 (2) | 1 (1)
Injection site pruritus (General disorders) | 4 (8) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Retinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraocular pressure (IOP) increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscles spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 1 (2)
Parasthesia (Nervous system disorders) | 1 (2) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nipple swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Orapharyngeal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Visual acuity decreased (II) (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 2 (5) | 0 (0)
Injection site pain (General disorders) | 5 (23) | 0 (0)
Injection site rash (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less